CLINICAL TRIAL: NCT02221895
Title: The Effect of Early (2-3 Week Postpartum) Versus Traditional (6-8 Week Postpartum) Follow-Up on Breastfeeding Rates at 6 Months
Brief Title: The Effect of Early Versus Traditional Follow-Up on Breastfeeding Rates at 6 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 214030
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy; Breastfeeding; Contraception; Cervical Cancer; Postpartum Depression
Keywords: postpartum appointment; breastfeeding; postpartum contraception; postpartum cervical cancer screening; postpartum depression screening
MeSH Terms: conditions — Breast Feeding; Uterine Cervical Neoplasms; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Follow-up (Experimental): Postpartum follow up appointment 2-3 weeks after delivery
  Interventions: Other: Postpartum follow up appointment 2-3 weeks after delivery
- Traditional Follow-up (Active Comparator): Postpartum follow up 6-8wk after delivery (current clinical standard)
  Interventions: Other: Postpartum follow up 6-8wk after delivery

INTERVENTIONS:
Other: Postpartum follow up appointment 2-3 weeks after delivery — experimental arm
  Arms: Early Follow-up
Other: Postpartum follow up 6-8wk after delivery — control arm
  Arms: Traditional Follow-up

SUMMARY:
The study's purpose is to determine if early (2-3 week) versus traditional (6-8 week) postpartum follow up is associated with a higher rate of breastfeeding at 6 months. The study's hypothesis is that follow up at 2-3 weeks postpartum is associated with a higher rate of breastfeeding 6 months postpartum.

DETAILED DESCRIPTION:
This study is a non-blinded randomized controlled trial with intent to treat analysis intended to determine whether early (2-3 weeks postpartum-experimental arm) versus traditional (6-8 weeks postpartum-control arm) follow up increases breastfeeding rates at 6 months' postpartum. For purposes of this study, breastfeeding will be defined as any breast milk produced by the mother and fed to her infant (whether by placing the infant to the breast or pumping/expressing milk and feeding it to the infant in another way). A literature search failed to identify any study that evaluated benefits or shortcomings of an exclusive short interval postpartum visit instead of the 6-8 week traditionally timed visit. Although there may be practical reasons to delay postpartum follow up until 6-8 weeks after delivery, there is no good data to support this, and it may remain the dominant practice due solely to convention. Recent expert opinion has suggested that earlier postpartum follow up may be more practical and provide an earlier or more convenient opportunity to provide assessment and education to postpartum women [9]. Earlier follow up may present a more timely opportunity to discuss family planning, breastfeeding, and screen for depression. Pierce CountyWomen/Infants/Children Program (WIC) data indicates a 34% breastfeeding rate in the military beneficiary population 6 months' postpartum (2012 data). Using a sample size of 166 in the exposure and non-exposure arms would allow for detection of a 50% increase in the outcome of the exposure arm using a two-sided test with α = 0.05 and β = 0.20. A 50% increase in the rate of breastfeeding 6 months' postpartum (from 34% to 51%) would be a clinically significant increase that approximates the Surgeon General's 2020 goal of a 60.6% rate of breastfeeding at 6 months. We assume at 30% dropout rate, and therefore, plan to recruit a total of 346 patients to the study.

Potential enrollees will be evaluated, recruited, and enrolled using the process described in 6.2.3(b). A screening and enrollment log will track all patients reviewed for eligibility whether or not they met inclusion/exclusion criteria and, if so, whether participation in the study was accepted or declined. Patients who agree to enroll will sign the required study consent and complete the breastfeeding attrition prediction tool (BAPT). With the subject's assistance, the enrolling investigator will complete the demographic sheet. Once these items are complete, randomization will occur. Randomization will be via computer-generated block randomization with block sizes of six. Randomization and blocking will be performed using the RAND function in Excel. Randomization will be performed by the study's collaborating staff, who will have no direct contact with the potential subjects. Treatment "A" will represent follow up 2-3 weeks postpartum. Treatment "B" will represent follow up at 6-8 weeks postpartum. The randomized assignments denoted as either "Treatment A: 2-3 week follow up" or "Treatment B: 6-8 week follow up" will be placed on a card within sequentially numbered, sealed, opaque envelopes by the collaborating staff. The randomization process, card, and envelope preparation will all be completed by the collaborating staff without any involvement of the study investigators. These sequentially numbered and sealed envelopes will be secured on Labor and Delivery until the study investigator allocates an envelope to the enrollee. Once a patient agrees to enrollment, the required demographic and screening tools are completed and the study consent form signed, the box containing the sequentially numbered and sealed envelopes will be opened by the study investigator and the patient will be given the next envelope in the sequence. Prior to opening the envelope, the study investigator will denote on the enrollment log the date of subject enrollment and the sequence number of the envelope assigned to the subject. The envelope number assigned to the subject will be their study number. The subject will then open the assigned envelope to determine their treatment assignment, and the study investigator will denote the study arm assignment on the enrollment log.

Once assigned to a treatment arm, the screening and enrollment log designating treatment assignments will be used to coordinate with the clerk in the Ob/Gyn Clinic, who will contact the subject to schedule postpartum follow up at the allotted interval. The scheduled appointments will be with providers (nurse practitioners and nurse midwives) not associated with the study. At the postpartum visit, the subject will complete and return the postpartum questionnaire, along with the Edinburgh perinatal depression screen, which is standard screening completed by all postpartum patients. Subjects demonstrating an elevated depression screen will be followed and assessed according to previously approved departmental protocol (MAMC Perinatal Screening Program Algorithm). Subjects who fail to show up at the assigned follow up interval will be included in the 6-month postpartum assessment. Subjects who return for follow up at intervals outside their assigned appointment interval will also be contacted for the 6- month follow up and included in their originally assigned group for data analysis (intent-to-treat).

When the patient is 5-6 months' postpartum, a study investigator will telephonically contact the subject to obtain answers to the 6-month postpartum questionnaire. The questionnaire will be reviewed by standardized script.

A multitude of factors influence breastfeeding success for mothers choosing to breastfeed. Some of these factors include prior breastfeeding experience, maternal and fetal medical complications, social support, attitudes, education, age, race, and other demographic factors, as well as maternal-fetal proximity within the immediate postpartum period. To minimize potential confounders and bias, we aim to enroll only primiparous mothers, as these mothers are unlikely to have prior breastfeeding experience. Demographic information collected will be used to perform subset analyses and evaluate the homogeneity of the two study groups. The standardized assessment tools will be used to characterize maternal attitudes and support for breastfeeding and will also be used for subset analysis. Some neonates are unable to be with their mother immediately after birth due to a variety of issues that may warrant observation in the Neonatal Intensive Care Unit (NICU) or, in some cases, due to maternal illness. We will also exclude mothers whose infants are not rooming-in with them continuously for the first 48 hours postpartum, as this may pose a potential barrier to initiating breastfeeding. To ensure the study is generalizable, we will include mothers with spontaneous or operative deliveries, as well as cesarean deliveries, which constitute approximately 16% (nulliparous term singleton vertex cesarean birth rate at our facility in 2012) of primiparous births at our facility, as long as the other inclusion/exclusion criteria are met. Additionally, some patients may present for enhanced follow up (in the case of a complicated delivery or postpartum complication) or acute visits within the first 8 weeks' postpartum. These visits represent other opportunities outside the typical postpartum follow up appointment for mothers to seek evaluation for breastfeeding support or other concerns. We will collect data on the number and type of scheduled and unscheduled provider encounters that occur within our medical system outside of the scheduled postpartum follow up appointment. Furthermore, some subjects may fail to follow up at the assigned interval. Data analysis will be via an intent-to-treat, therefore, subjects assigned to one arm or the other who either fail to follow up at the assigned interval or follow up more frequently will still be evaluated and assessed for the primary outcome.

1. Describe what will happen on this study that is EXPERIMENTAL: Subjects in the experimental arm (2-3 week postpartum follow up) will have their postpartum appointment at an earlier interval that what is current considered the standard of care. All study participants will complete the BAPT. Demographic data will be obtained for each subject prior to their discharge. All subjects will also complete a standardized postpartum questionnaire at their scheduled postpartum visit (either 2-3 weeks or 6-8 weeks depending on their arm of the study). All subjects will have a 6-month follow up via a standardized/scripted phone survey.
2. Describe what will happen on this study that is STANDARD of CARE: The control arm of the trial will be assigned to the traditional 6-8 week postpartum visit. All study subjects will receive postpartum follow up care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above at time of delivery
* Delivery of live born infant at estimated gestational age (EGA) ≥37wk
* Postpartum primiparous patients within the first 48 hours after delivery
* Patient intent to breastfeed
* Breastfeeding initiated within the first 48 hours of delivery and/or prior to hospital discharge (whichever occurs first)
* Infant is continuously rooming in with mother from the time of delivery
* English-speaking
* Able to read and complete surveys
* No anticipated discharge from military system, Tricare benefits, or move planned in the upcoming 6 months
* Willing to render informed consent

Exclusion Criteria:

* Patients delivered by the Family Medicine Department (relatively small number in our population who are not followed postpartum by the Department of Obstetrics and Gynecology)
* Any condition deemed by patient provider to be an absolute contraindication to breastfeeding
* Maternal HIV/AIDS
* Planned use of radioactive or chemotherapeutic medications or medication for other medical problems which is contraindicated for delivery
* Known fetal factor that would impair breastfeeding
* Fetal mid-facial defects
* Known fetal chromosomal abnormality
* Known fetal conditioning resulting in fetal hypotonia
* Labor and Delivery complications
* Maternal separation from infant during the first 48 hours postpartum (such as maternal ICU admission, infant NICU admission)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2014-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
breastfeeding | 5-6 months postpartum
  Breastfeeding is defined, for purposes of this study, as any breast milk produced by the mother and fed to the infant (by placing the infant to the breast or by pumping or manually expressing and feeding to the infant by other means). Nominal/categorical assessment (breastfeeding to any degree: yes or no) of breastfeeding will be used to determine the primary outcome.

SECONDARY OUTCOMES:
breastfeeding | 5-6 months postpartum
  Subset analysis of primary outcome using additional nominal characterization (breastfeeding only with no other foods/water, breastfeeding with some table foods, breastfeeding and formula feeding with or without some table foods, formula feeding with or without some table foods, formula only).
Contraception | up to 6 months after delivery
  Choice, use, prescription for contraception in the 6 months postpartum period.
Depression screen | up to 8wk postpartum
  Score of Edinburgh depression screen at time of postpartum encounter
Appointment utilization | 8wk postpartum
  Total number of appointments in the 8 weeks after delivery
BAPT | within 48hr of enrollment
  use of the BAPT screening tool to predict breastfeeding attrition
Cervical cancer screening | up to 8wk postpartum
  number of patients who had a pelvic examination at the time of their postpartum appointment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Abbott, MD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abbott JL, Carty JR, Hemman E, Batig AL. Effect of Follow-Up Intervals on Breastfeeding Rates 5-6 Months Postpartum: A Randomized Controlled Trial. Breastfeed Med. 2019 Jan/Feb;14(1):22-32. doi: 10.1089/bfm.2018.0071. Epub 2018 Nov 9. PMID 30412416